CLINICAL TRIAL: NCT05839249
Title: The Impact of Covid 19 Pandemic on Ureteric Stents Complications.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Mostafa AbdelRazek, Assistant Professor of Urology, South Valley University
Other Study IDs: SVU/MED/URO016/2.23.4.539
Record Dates: First submitted 2023-04-28; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Determine Effect of Urological Malpractice During Covid 19 on Patient Complications
Keywords: urological stents , COVID19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: JJ urological stents — recording complications of JJ stents during COVID19 pandemics

SUMMARY:
The pandemic of coronavirus disease 2019 (COVID-19) has serious implications on urology practice and raises particular questions for urologists about the management of different conditions. It was recommended to cancel most of the elective urological surgeries. (1) The least invasive intervention modalities that can be completed in local or regional anesthesia will serve the best interest of patients and urologists. 10 14 Endoscopic surgery is considered relatively safe.(2) After end of pandemic we facing complication of this era, one of most common complication was JJ stents complications as most of patient and doctors prefers to defer most of elective management by just JJ insertion and postpone definitive treatment. (3) In this study we discuss retrospectively the complication of JJ stenting during Covid 19 pandemic.

DETAILED DESCRIPTION:
Type of the study: retrospective clinical study

* Study Setting: Qena University Hospital 3- Study subjects:

  a. Inclusion criteria: all patients performing JJ stent placement during Covid 19 pandemics b. Exclusion criteria: Patients refuse to participate in this study c. Sample Size Calculation: all patients performing JJ stent placement from March 2020 to December 2021
* Study tools (in detail, e.g., lab methods, instruments, steps, chemicals, …):

  * Medical history
  * Complete physical examination.
  * All patents presented was investigated by

    1. Abdominal U.S
    2. Plain X Ray
    3. Non contrast CT
    4. Serum Creatinine
    5. Urine Analysis
* Research outcome measures:

  1. Primary (main): determine effect of urological malpractice during Covid 19 on patient complications
  2. Secondary (subsidiary): determine JJ stent complications during Covid 19 pandemics

ELIGIBILITY:
Inclusion Criteria:

* all patients performing JJ stent placement during Covid 19 pandemics

Exclusion Criteria:

* Patients refuse to participate in this study

Ages: 6 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patients performing JJ stent placement from January 2020 to December 2021
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-05-15 (Estimated)

PRIMARY OUTCOMES:
jj stents complications during covid 19 pandimics | 3 years
  determine effect of urological malpractice during Covid 19 on patient complications

CONTACTS AND LOCATIONS:
Locations (1):
- South Valley University, Qina, Qena Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No